CLINICAL TRIAL: NCT02620202
Title: Aiming Towards Evidence Based Interpretation of Cardiac Biomarkers in Patients Presenting With Chest Pain (WESTCOR Study)
Brief Title: Aiming Towards Evidence Based Interpretation of Cardiac Biomarkers in Patients Presenting With Chest Pain
Acronym: WESTCOR
Status: Terminated | Type: Observational
Why Stopped: It was no longer possible to include patients due to logistic challanges occuring during the Covid-19 pandemic
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/1365
Record Dates: First submitted 2015-10-12; First posted 2015-12-02 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2020-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Troponin; Myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Full blood, Serum samples, EDTA plasma, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The main aim of the WESTCOR study is to

* investigate the ability of two high sensitive cardiac troponin (hs-cTn) assays to diagnose acute coronary syndrome and predict prognosis in different patient populations (e.g. gender, age and co-morbidity)
* to validate the suggested 1 hour protocol for rule in and rule out of acute coronary syndrome for two hs-cTn assays in an unselected chest pain population
* to investigate different biomarkers ability to predict long term prognosis after hospitalization for chest pain

DETAILED DESCRIPTION:
The WESTCOR-study will include patients presenting to the Emergency Department of Haukeland University Hospital and Stavanger University Hospital with symptoms indicative of acute coronary syndrome. 1500 patients will be included at Haukeland University Hospital and 400 at Stavanger University Hospital. The two locations use different high sensitive troponin assays (i.e. hs-cTnT and hs-cTnI (Abbott Diagnostics) for routine diagnostic of coronary syndrome.

1900 patients will be sampled and hs-cTnT or hs-cTnI (as applicable) will be measured at admission, after one (2/3 of the cohort), three hours and after 8-12 hours. Clinicians will be blinded to the results of the hs-cTn assay that is not used as routine assay locally. Final diagnosis will be made by two independent cardiologists based on all available clinical information and results of the routine tests. The ability to diagnose or exclude MI ACS, and MACE at different sampling points in different patient populations will be compared for different biomarkers. 1500 patients will have a sample 1 hour after admission. The clinicians will be blinded to the results of this sample (both hs-cTn assays). The ability of the one-hour sample to diagnose or exclude myocardial infraction (MI), ACS and MACE will be compared between biomarkers.

All patients will be invited to take a follow-up sample 3 months after discharge.

The patients will further be followed for 1-5 years through national registers and the prognostic value of hs-cTn concentrations and dynamics as well as other biomarkers, will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Emergency Department with a clinical suspicion of acute coronary syndrome i.e. chest pain or pain radiating down the arms, the back, into the jaw, throat or into the lower teeth. Chest pain must not be the most dominant symptom but may or may not be combined with e.g. dyspnea, nausea, anxiousness or palpitations.
* Age >= 18 years

Exclusion Criteria:

* ST elevation MI
* Age < 18 years
* Patients not able to give informed consent
* Patients suffering from terminal illness (life expectance < 1 month)
* Patients already included in the study
* Patients who have been stabilized at local hospitals and are referred for second opinion e.g. coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Emergency Department at Haukeland University Hospital or Stavanger University Hospital with symptoms indicative of acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with chest pain that are diagnosed with acute coronary syndrome based on troponin concentrations | 1-3 hours
  Stratified according to gender, age and co-morbidities

OTHER OUTCOMES:
Number of patients with chest pain that are diagnosed with NSTEMI based on troponin concentration | 1-3 hours
  Stratified according to gender, age and co-morbidities
Total mortality | 5 years
  Patients will be followed for 1-5 years through national registers
The incidence of major cardiovascular events (MACE) defined as (composite endpoint including MI, UAP, stable angina (requiring hospitalization), revascularization, stroke, heart failure and cardiac arrhythmias) | 5 years
  Patients will be followed for 1-5 years through national registers
Cardiovascular mortality | 5 years
  Patients will be followed for 1-5 years through national registers
The incidence of major coronary events defined as (composite endpoint including MI, UAP, stable angina (requiring hospitalization), revascularization) | 5 years
  Patients will be followed for 1-5 years through national registers

CONTACTS AND LOCATIONS:
Overall Officials: Kristin M Aakre, MD, PhD, Principal Investigator — Laboratory of Clinical Biochemistry, Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger

REFERENCES:
- [Derived] Saeed N, Restan IZ, Steiro OT, Tjora HL, Langorgen J, Skadberg O, Mjelva OR, Bonarjee VVS, Bjorneklett RO, Steinsvik T, Vikenes K, Omland T, Apple FS, Jaffe AS, Mills NL, Collinson PO, Kavsak PA, Aakre KM. Analytical Error of Cardiac Troponin and Impact on the Performance of Accelerated Diagnostic Protocols in Patients with Acute Chest Pain. Clin Chem. 2025 Dec 2;71(12):1243-1256. doi: 10.1093/clinchem/hvaf116. PMID 41092105
- [Derived] Saeed N, Steiro OT, Langorgen J, Tjora HL, Bjorneklett RO, Skadberg O, Bonarjee VVS, Mjelva OR, Norekval TM, Steinsvik T, Vikenes K, Omland T, Aakre KM. Diagnosing Myocardial Injury in an Acute Chest Pain Cohort; Long-Term Prognostic Implications of Cardiac Troponin T and I. Clin Chem. 2024 Oct 3;70(10):1241-1255. doi: 10.1093/clinchem/hvae110. PMID 39119917
- [Derived] Saeed N, Norekval TM, Steiro OT, Tjora HL, Langorgen J, Bjorneklett RO, Skadberg O, Bonarjee VVS, Mjelva OR, Omland T, Vikenes K, Aakre KM. Predictors of long-term symptom burden and quality of life in patients hospitalised with chest pain: a prospective observational study. BMJ Open. 2022 Jul 13;12(7):e062302. doi: 10.1136/bmjopen-2022-062302. PMID 35831040
- [Derived] Steiro OT, Aakre KM, Tjora HL, Bjorneklett RO, Skadberg O, Bonarjee VVS, Mjelva OR, Omland T, Vikenes K, Langorgen J. Association between symptoms and risk of non-ST segment elevation myocardial infarction according to age and sex in patients admitted to the emergency department with suspected acute coronary syndrome: a single-centre retrospective cohort study. BMJ Open. 2022 May 12;12(5):e054185. doi: 10.1136/bmjopen-2021-054185. PMID 35551077